CLINICAL TRIAL: NCT00017121
Title: Dose Finding Study of Aerosolized GM-CSF in the Treatment of Metastatic Melanoma to the Lung
Brief Title: Inhaled Sargramostim in Treating Patients With Melanoma Metastatic to the Lung
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0071; NCI-2012-02385 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000068654 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Melanoma (Skin); Metastatic Cancer
Keywords: stage IV melanoma; recurrent melanoma; lung metastases
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sargramostim (Experimental): Patients receive aerosolized sargramostim (GM-CSF) twice a day on days 1-7 and 15-21. Treatment repeats every 28 days for 2 courses. Patients with no disease progression after completion of course 2 may continue on treatment until disease progression. Patients are grouped to 1 of 2 dose-escalation regimens (part A vs B).
  After completion of study therapy, patients are followed at 3 months, every 2 months for 1 year, and then every 3-4 months for 5 years.
  Interventions: Biological: sargramostim

INTERVENTIONS:
Biological: sargramostim

SUMMARY:
RATIONALE: Inhaling sargramostim may interfere with the growth of tumor cells and may be an effective treatment for melanoma that has spread to the lung.

PURPOSE: This phase I trial is studying the side effects and best dose of inhaled sargramostim in treating patients with melanoma that is metastatic to the lung.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine immunomodulatory effects of aerosolized sargramostim (GM-CSF) in patients with metastatic melanoma to the lung (part A).
* Determine toxicity profile of this therapy, in terms of pulmonary and hematologic toxicity, in these patients.
* Determine, preliminarily, the therapeutic effects of this therapy, in terms of progression-free survival, overall survival, and objective response rate, in these patients.
* Determine the maximum tolerated dose of GM-CSF in these patients (part B).

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive aerosolized sargramostim (GM-CSF) twice a day on days 1-7 and 15-21. Treatment repeats every 28 days for 2 courses. Patients with no disease progression after completion of course 2 may continue on treatment until disease progression. Patients are grouped to 1 of 2 dose-escalation regimens (part A vs B).

* Part A: Cohorts of 5-10 patients receive escalating doses of GM-CSF until the optimal immunostimulatory dose (ISD) is determined. The optimal ISD is defined as the dose at which at least 7 of 10 patients experience immunostimulation. Once the optimal ISD is determined, 10 patients receive aerosolized GM-CSF at a dose halfway between the optimal ISD and the preceding dose. Dose escalation is discontinued if at least 2 of 5 or at least 4 of 10 patients on a particular dose level experience dose-limiting toxicity.
* Part B: Cohorts of 3-6 patients receive escalating doses of GM-CSF until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

After completion of study therapy, patients are followed at 3 months, every 2 months for 1 year, and then every 3-4 months for 5 years.

PROJECTED ACCRUAL: A total of 85 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma to the lung for which no known standard therapy exists
* At least 1 unidimensionally measurable lesion
* HLA-A2 positive (part A patients only)
* Previously treated CNS metastases allowed provided there is no evidence of disease progression within the past 3 months

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 8.0 g/dL

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST no greater than 3 times ULN

Renal:

* Creatinine no greater than 2.5 times ULN

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Pulmonary:

* No pulmonary disease requiring concurrent active therapy (e.g., supplemental oxygen or bronchodilator)
* FEV_1 at least 65% of predicted and at least 1.5 L

Immunologic:

* No known immunodeficiency state
* No known autoimmune disease
* No uncontrolled infection

Other:

* No active psychotic disorder requiring pharmacotherapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 2 weeks since prior biologic therapy
* More than 2 weeks since prior immunotherapy
* More than 4 weeks since prior filgrastim (G-CSF) or sargramostim (GM-CSF)
* No other concurrent biologic therapy or immunotherapy
* No concurrent G-CSF
* No concurrent GM-CSF other than study drug

Chemotherapy:

* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No concurrent chemotherapy

Endocrine therapy:

* More than 2 weeks since prior corticosteroids
* No concurrent glucocorticosteroids

Radiotherapy:

* More than 2 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* More than 7 days since prior parenteral antibiotics
* No concurrent parenteral antibiotics
* No concurrent immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Up to 6 years

SECONDARY OUTCOMES:
Progression-free survival | Up to 6 years
Overall survival | Up to 6 years
Objective response rate | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, MD, PhD, Study Chair — Mayo Clinic
Locations (87):
- United States (87):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA at Maplewood Cancer Center, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Hematology-Oncology Associates of Fredericksburg, Incorporated, Fredericksburg, Virginia

REFERENCES:
- [Result] Markovic SN, Suman VJ, Nevala WK, Geeraerts L, Creagan ET, Erickson LA, Rowland KM Jr, Morton RF, Horvath WL, Pittelkow MR. A dose-escalation study of aerosolized sargramostim in the treatment of metastatic melanoma: an NCCTG Study. Am J Clin Oncol. 2008 Dec;31(6):573-9. doi: 10.1097/COC.0b013e318173a536. PMID 19060590
- [Result] Markovic SN, Suman VJ, Schaefer P, et al.: Aerosolized sargramostim for the treatment of metastatic melanoma to the lungs. [Abstract] J Clin Oncol 25 (Suppl 18): A-8565, 488s, 2007.